CLINICAL TRIAL: NCT01810263
Title: The Efficacy of Intensive Nutritional Supplement in Patient With Stroke: a Prospective Randomized Controlled Trial
Brief Title: The Efficacy of Intensive Nutritional Supplement in Patient With Stroke
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The study does not seem to provide benefits to patients.
Sponsor: Seoul National University Bundang Hospital (Other)
Collaborators: Myongji Hospital (Other)
Responsible Party: Principal Investigator, Nam-Jong Paik, professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B-1112-069-007
Record Dates: First submitted 2013-02-01; First posted 2013-03-13 (Estimated); Results first posted 2015-07-02 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-07

CONDITIONS: Stroke; Malnutrition
Keywords: stroke; malnutrition; high protein
MeSH Terms: conditions — Stroke; Malnutrition

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- high protein supplement (Experimental): high protein supplement given
  Interventions: Dietary Supplement: high protein supplement
- Control (No Intervention): no intervention

INTERVENTIONS:
Dietary Supplement: high protein supplement — Dietary Supplement: high protein supplement
  Other Names: Intensive Nutritional Supplement group
  Arms: high protein supplement

SUMMARY:
The aim of this prospective randomized controlled study is to demonstrate the efficacy of Intensive Nutritional Supplement in Patient with Stroke.

DETAILED DESCRIPTION:
Elderly patients, including those who have had a stroke, are more at risk of undernutrition than other groups because of reduced nutritional reserves, prolonged hospital stay and increased demands of repeated ill-health. Stroke may compound these problems because of physical and mental incapacity, problems with perception and communication, and swallowing disorders. The full extent of undernutrition and its independent contribution to stroke outcome is not presently known. It is also not known whether it can be corrected, and whether doing so would improve the outcome. The aim of this study is therefore to describe the efficacy of Intensive Nutritional Supplement in Patient with Stroke.

ELIGIBILITY:
Inclusion Criteria:

* 1 st onset stroke patient
* MRI confirms his/her stroke
* more than 2.5% weight los within 2 weeks
* initial serum albumin < 35 g/l
* BMI < 18.5
* more than MMSE 10
* medically stable

Exclusion Criteria:

* recurrent stroke patient
* malabsorption patient
* terminal cancer

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nam-Jong Paik, MD, PhD, Principal Investigator — Department of Rehabilitation Medicine, Seoul National University College of Medicine, Seoul National University Bundang Hospital, Seongnam, Korea
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Korea, Gyeonggi-do, South Korea

REFERENCES:
- [Background] Gariballa SE, Parker SG, Taub N, Castleden M. Nutritional status of hospitalized acute stroke patients. Br J Nutr. 1998 Jun;79(6):481-7. doi: 10.1079/bjn19980085. PMID 9771334
- [Background] Axelsson K, Asplund K, Norberg A, Alafuzoff I. Nutritional status in patients with acute stroke. Acta Med Scand. 1988;224(3):217-24. doi: 10.1111/j.0954-6820.1988.tb19364.x. PMID 3239449
- [Derived] Sakai K, Niimi M, Momosaki R, Hoshino E, Yoneoka D, Nakayama E, Masuoka K, Maeda T, Takahashi N, Sakata N. Nutritional therapy for reducing disability and improving activities of daily living in people after stroke. Cochrane Database Syst Rev. 2024 Aug 15;8(8):CD014852. doi: 10.1002/14651858.CD014852.pub2. PMID 39145517

RESULTS

PARTICIPANT FLOW:
Recruitment Details: * first ever stroke
  * MRI confirms his/her stroke
  * weight loss over 2.5% within 2 weeks after the stroke onset
  * MMSE >= 10
  * medically stable
Groups:
- High Protein Supplement: Patients in the both groups keep on routine diet in the hospital All the patients in the High Protein Supplement group were provided additional calories of Nucare(High protein fluid diet, 200kcal/200ml/1 can. Dasang, Seoul, Korea) three times a day.
  (As a result, additional calories are 600kcal a day)
- Control: Patients in the both groups keep on routine diet in the hospital. No additional calories are provided.
Period: Overall Study
Arm/Group | High Protein Supplement | Control
Started | 16 | 18
Completed | 8 (2014 July) | 11
Not Completed | 8 | 7
Not completed — Lost to Follow-up | 8 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Protein Supplement | Control | Total
Number analyzed (Participants) | 16 | 18 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (16.0) | 65.8 (14.3) | 64.4 (15.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 7 | 11 | 18
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 16 | 18 | 34

OUTCOME MEASURES:

1. Primary Outcome: Modified Barthel Index (MBI) Score at 6 Months
Description: Scale range: 0-100 (higher values represent a better outcome)
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | High Protein Supplement | Control
Number analyzed (Participants) | 16 | 18
units on a scale | 23.3 (2.7) | 21.9 (2.7)

2. Secondary Outcome: Chemical Laboratory Findings
Time Frame: 6 months
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Body Mass Index
Time Frame: 6 months
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Triceps Skin Fold Thickness
Time Frame: 6 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Subjective Global Assessment
Time Frame: 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Description: Serious and other non-serious adverse events were not reported.
Arm/Group | High Protein Supplement | Control
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/18
Other Adverse Events (participants affected / at risk) | 0/16 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No